CLINICAL TRIAL: NCT00197184
Title: Evaluate the Persistence of Immune Response of GSK Biologicals' Twinrix™ Vaccine, Administered According to a 0,6 Month Schedule and a 0,1,6 Month Schedule, in Healthy Children Aged Between 1-11 Years at the Time of First Vaccine Dose
Brief Title: Long Term Follow-up Study at Years 2, 3, 4 and 5 Where 2 Dosing Schedules of the Combined Hepatitis A and B Vaccine Were Compared
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 208127/132 (EXT Y2); 208127/133 (EXT Y3) (Other: GSK); 208127/134 (EXT Y4) (Other: GSK); 208127/137 (EXT Y5) (Other: GSK); NCT00787449 (obsolete NCT alias)
Record Dates: First submitted 2005-09-15; First posted 2005-09-20 (Estimated); Results first posted 2009-06-04 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2016-10

CONDITIONS: Hepatitis B; Hepatitis A
Keywords: Combined hepatitis A and B vaccine; Twinrix™
MeSH Terms: conditions — Hepatitis B; Hepatitis A

ARMS (2):
- Twinrix Junior (Experimental): Subjects previously received 3 doses of combined hepatitis A / hepatitis B vaccine (junior formulation).
  Interventions: Biological: Twinrix™ Junior
- Twinrix Adult (Active Comparator): Subjects previously received 2 doses of combined hepatitis A / hepatitis B vaccine (adult formulation).
  Interventions: Biological: Twinrix™ Adult

INTERVENTIONS:
Biological: Twinrix™ Adult — Intramuscular injection in the left deltoid, 2 doses, Adult formulation in primary study.
  Other Names: Combined hepatitis A and B vaccine
  Arms: Twinrix Adult
Biological: Twinrix™ Junior — Intramuscular injection in the left deltoid, 3 doses, junior formulation in primary study.
  Other Names: Combined hepatitis A and B vaccine
  Arms: Twinrix Junior

SUMMARY:
To evaluate the persistence of anti-hepatitis A virus (HAV) and anti-hepatitis B surface antigen (HBs) antibodies up to 2, 3, 4 and 5 years after administration of the first dose of the study vaccine.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

DETAILED DESCRIPTION:
Open, randomised, self-contained, multicentric, multinational, long-term antibody persistence studies. Immune persistence was compared between subjects who received either two dose or three doses of GSK Biologicals combined hepatitis A and hepatitis B vaccine. The long-term follow-up studies involved taking blood samples at approximately 2, 3, 4 and 5 years after the primary vaccination of combined hepatitis A and B vaccine to assess antibody persistence. No additional subjects will be recruited during the long term follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Participation in primary study
* Written informed consent obtained before each long term follow up visit.

Ages: 3 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 276 (Actual)
Dates: Start 2003-11-01; Primary Completion 2004-03-10 (Actual); Study Completion 2004-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- Australia (2):
  - GSK Investigational Site, North Adelaide, South Australia
  - GSK Investigational Site, Carlton, Victoria
- GSK Investigational Site, Brussels, Belgium
- Spain (4):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Blanes (Girona)
  - GSK Investigational Site, Cerdanyola Del Vallés / Barcelona
  - GSK Investigational Site, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Marshall H, Nolan T, Diez Domingo J, Rombo L, Sokal EM, Mares J, Casanovas JM, Kuriyakose S, Leyssen M, Jacquet JM. Long-term (5-year) antibody persistence following two- and three-dose regimens of a combined hepatitis A and B vaccine in children aged 1-11 years. Vaccine. 2010 Jun 17;28(27):4411-5. doi: 10.1016/j.vaccine.2010.04.040. Epub 2010 Apr 29. PMID 20434544
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 208127/132 (EXT Y2) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 208127/132 (EXT Y2) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 208127/132 (EXT Y2) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 208127/132 (EXT Y2) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 208127/132 (EXT Y2) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 208127/132 (EXT Y2) — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register. The results of this study 208127/132 are summarised with studies 208122/133, 208127/134 and 208127/137 on the GSK Clinical Study Register.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Twinrix Adult | Twinrix Junior
Started | 139 | 137
Completed | 139 | 137
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Twinrix Adult | Twinrix Junior | Total
Number analyzed (Participants) | 139 | 137 | 276
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.6 (2.97) | 11.2 (3.11) | 11.4 (3.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 64 | 123
  Male | 80 | 73 | 153

OUTCOME MEASURES:

1. Primary Outcome: Anti-hepatitis A (HAV) Antibody Concentrations
Description: Geometric mean concentration for anti-HAV antibodies expressed as Milli-International Units per milliliter (mIU/mL)
Time Frame: Year 2 (Month 24), Year 3 (Month 36), Year 4 (Month 48) and Year 5 (Month 60)
Population: Analysis was performed on the Long Term According to Protocol cohort for analysis of immunogenicity (LT ATP immunogenicity cohort) which included all subjects that complied with the protocol and for whom data concerning immunogenicity endpoint measures were available for the particular time point measured.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Twinrix Adult | Twinrix Junior
Number analyzed (Participants) | 129 | 119
mIU/mL
  At year 2: number analyzed (Participants) | 107 | 94
  At year 2 | 1122.2 [937.7 to 1343.0] | 1377.8 [1114.0 to 1704.2]
  At year 3 | 998.6 [845.8 to 1178.9] | 1347.1 [1145.1 to 1584.8]
  At year 4: number analyzed (Participants) | 115 | 105
  At year 4 | 737.5 [623.6 to 872.3] | 915.9 [774.0 to 1084.0]
  At year 5: number analyzed (Participants) | 103 | 101
  At year 5 | 576.8 [473.6 to 702.5] | 698.4 [585.1 to 833.7]

2. Primary Outcome: Anti-hepatitis B (HBs) Antibody Concentrations
Description: Geometric mean concentration for anti-HBs antibodies expressed as Milli-International Units per milliliter (mIU/mL).
Time Frame: Year 2 (Month 24), Year 3 (Month 36), Year 4 (Month 48) and Year 5 (Month 60)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Twinrix Adult | Twinrix Junior
Number analyzed (Participants) | 129 | 119
mIU/mL
  At year 2: number analyzed (Participants) | 107 | 94
  At year 2 | 479.9 [356.6 to 646.0] | 830.6 [609.5 to 1131.9]
  At year 3 | 325.1 [244.7 to 431.8] | 695.1 [516.5 to 935.5]
  At year 4: number analyzed (Participants) | 115 | 105
  At year 4 | 270.2 [201.0 to 363.3] | 519.7 [378.5 to 713.6]
  At year 5: number analyzed (Participants) | 102 | 100
  At year 5 | 150.2 [110.5 to 204.3] | 283.7 [208.6 to 386.0]

3. Primary Outcome: Anti-HAV Antibody Concentrations in Subjects Receiving the Additional Vaccine Dose.
Description: Any subjects becoming seronegative for anti-HAV antibodies (i.e. titres < 15 mIU/ml) at any long term time point, were to receive an additional vaccine dose administered between 6 to 12 months after Year 5 time point.
Time Frame: Before and one month after additional vaccination
Population: None of the subjects became seronegative for anti-HAV antibodies during the Year 2 to Year 5 long term follow-up. Hence none of the subjects received an additional Havrix dose.
Arm/Group | Twinrix Adult | Twinrix Junior
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Anti-HBs Antibody Concentrations in Subjects Receiving the Additional Vaccine Dose.
Description: Subjects losing seroprotective anti-HBs antibody titres (i.e. titres < 10 mIU/ml) at any long term time point, received an Engerix challenge dose. The table presents the geometric mean concentrations for anti-HBs antibodies, expressed as Milli-International Units per milliliter (mIU/mL).
Time Frame: Before and One month after additional vaccination
Population: Analysis was performed on the Total vaccinated cohort for the challenge dose, including all subjects who received an additional vaccine dose between 6 to 12 months after year 5.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Twinrix Adult | Twinrix Junior
Number analyzed (Participants) | 11 | 5
mIU/mL
  Before vaccination: number analyzed (Participants) | 6 | 1
  Before vaccination | 4.9 [2.1 to 11.1] | 2.4 [0.9 to 6.5]
  Post vaccination | 521.3 [158.2 to 1718.1] | 509.7 [173.5 to 1497.9]

5. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs) Determined by the Investigator to Have a Causal Relationship to Primary Vaccination or Due to Lack of Vaccine Efficacy.
Description: A serious adverse event (SAE) is any untoward medical occurrence that:
  results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study subject, or may evolve into one of the outcomes listed above.
Time Frame: From last study visit of the primary study up to Year 5 long term follow-up
Population: The analysis was performed on the Long term Total vaccinated cohort wich included all subjects who returned at a specified follow-up study
Measure: Count of Participants; unit: Participants
Arm/Group | Twinrix Adult | Twinrix Junior
Number analyzed (Participants) | 139 | 137
Participants | 0 | 0

6. Secondary Outcome: Number of Subjects Receiving an Additional Vaccine Dose and Reporting Solicited Local Symptoms
Description: Solicited local symptoms assessed include pain, redness and swelling at the vaccine injection site.
  Any= regardless of intensity grade; Grade 3 Pain= spontaneously painful
Time Frame: during the 4-day follow-up period after additional vaccination
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Twinrix Adult | Twinrix Junior
Number analyzed (Participants) | 11 | 5
Participants
  Pain, any | 6 | 0
  Pain, grade 3 | 0 | 0
  Redness, any | 1 | 0
  Redness, >20mm | 0 | 0
  Swelling, any | 0 | 0
  Swelling, >20mm | 0 | 0

7. Secondary Outcome: Number of Subjects Receiving an Additional Vaccine Dose and Reporting Solicited General Symptoms.
Description: Solicited general symptoms assessed include fatigue, fever, gastrointestinal symptoms and headache.
  Any= regardless of intensity grade or relationship to vaccination; grade 3= prevented normal activity; Related= considered by the investigator to be causally related to the vaccination
Time Frame: During the 4-day follow-up period after additional vaccination
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Twinrix Adult | Twinrix Junior
Number analyzed (Participants) | 11 | 5
Participants
  Fatigue, any | 3 | 0
  Fatigue, grade 3 | 0 | 0
  Fatigue, related | 3 | 0
  Fever (axillary), ≥37°C | 0 | 0
  Fever (axillary), >39.5°C | 0 | 0
  Fever (axillary), related | 0 | 0
  Gastrointestinal, any | 2 | 0
  Gastrointestinal, grade 3 | 0 | 0
  Gastrointestinal, related | 2 | 0
  Headache, any | 4 | 0
  Headache, grade 3 | 0 | 0
  Headache, related | 4 | 0

8. Secondary Outcome: Number of Subjects Receiving an Additional Vaccine Dose and Reporting Unsolicited Adverse Events (AEs).
Description: An Adverse Event is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: During the 30-day follow-up period after additional vaccination.
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Twinrix Adult | Twinrix Junior
Number analyzed (Participants) | 11 | 5
Participants | 2 | 0

9. Secondary Outcome: Number of Subjects Receiving an Additional Vaccine Dose and Reporting Any Serious Adverse Events
Description: as for outcome 5
Time Frame: At least one month after additional vaccination
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Twinrix Adult | Twinrix Junior
Number analyzed (Participants) | 11 | 5
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited symtoms: During the 4-day (Day 0-3) follow-up period after the additional vaccination. Unsolicited AEs: During the 31-day (Day 0-30) period after the additional vaccination; SAEs: During the entire study period
Description: Solicited and unsolicited symptoms were collected on the Total vaccinated cohort for the challenge dose for subjects who received the additional vaccine dose after the Year 5; SAEs were collected on the Long term Total vaccinated cohort throughout the study period.
Arm/Group | Twinrix Adult | Twinrix Junior
Serious Adverse Events (participants affected / at risk) | 0/139 | 0/137
Other Adverse Events (participants affected / at risk) | 7/11 | 0/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Twinrix Adult (N=11) | Twinrix Junior (N=5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Syncope vasovagal (Nervous system disorders) | 1 | 0
Balanitis (Reproductive system and breast disorders) | 1 | 0
Redness at the injection site (General disorders) | 1 | 0
Pain at the injection site (General disorders) | 6 | 0
Fatigue (General disorders) | 3 | 0
Gastrointestinal disorder (General disorders) | 2 | 0
Headache (General disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.